CLINICAL TRIAL: NCT02051959
Title: Long-Term Treatment of Patients Experiencing Phantom Limb Pain With Transcranial Direct Current Stimulation (tDCS)
Brief Title: Long-term Effects of Transcranial Direct Current Stimulation (tDCS) on Patients With Phantom Limb Pain (PLP)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Signing a contract with the company owning the equipment
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Itzhak Siev-Ner, Head of The Department of Orthopedic Rehabilitation, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-13-0733-IS-CTIL
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Phantom Limb Pain
Keywords: Phantom Limb Pain; Transcranial Direct Current Stimulation; Amputation; Diabetes Mellitus
MeSH Terms: conditions — Phantom Limb; Diabetes Mellitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Crossover 1a: anodal stimulation of M1 + sham (Active Comparator): 6 amputees will undergo 8 active treatments of 20 min 2mA anodal stimulation of M1 localized to the contralateral amputation area followed by 8 sham treatments.
  Total duration and frequency of treatments: 8 weeks, 2 sessions per week.
  Each session will last approximately one hour which will consist of:
  * EEG and pain measurements
  * 20 minutes of stimulation
  * EEG and pain measurements after completion of stimulation
  Interventions: Device: Anodal stimulation of M1 + sham
- Crossover 1b: sham + anodal stimulation of M1 (Active Comparator): 6 amputees will undergo 8 sham treatments followed by 8 active treatments of 20 min 2mA anodal stimulation of M1 localized to the contralateral amputation area.
  Total duration and frequency of treatments: 8 weeks, 2 sessions per week.
  Each session will last approximately one hour which will consist of:
  * EEG and pain measurements
  * 20 minutes of stimulation
  * EEG and pain measurements after completion of stimulation
  Interventions: Device: Sham + Anodal stimulation of M1
- Crossover 2a: cathodal stimulation of M1 + sham (Active Comparator): 6 amputees will undergo 8 active treatments of 20 min 2mA cathodal stimulation of M1 localized to the contralateral amputation area followed by 8 sham treatments.
  Total duration and frequency of treatments: 8 weeks, 2 sessions per week.
  Each session will last approximately one hour which will consist of:
  * EEG and pain measurements
  * 20 minutes of stimulation
  * EEG and pain measurements after completion of stimulation
  Interventions: Device: Cathodal stimulation of M1 + sham
- Crossover 2b: sham + cathodal stimulation of M1 (Active Comparator): 6 amputees will undergo 8 sham treatments followed by 8 active treatments of 20 min 2mA cathodal stimulation of M1 localized to the contralateral amputation area.
  Total duration and frequency of treatments: 8 weeks, 2 sessions per week.
  Each session will last approximately one hour which will consist of:
  * EEG and pain measurements
  * 20 minutes of stimulation
  * EEG and pain measurements after completion of stimulation
  Interventions: Device: Sham + Cathodal stimulation of M1

INTERVENTIONS:
Device: Anodal stimulation of M1 + sham — 8 active treatmments: 2mA anodal stimulation of M1 for 20 minutes (over the relevant cortex area) followed by 8 sham treatments.
  Other Names: tDCS
  Arms: Crossover 1a: anodal stimulation of M1 + sham
Device: Sham + Anodal stimulation of M1 — 8 sham treatments followed by 8 active treatmments: 2mA anodal stimulation of M1 for 20 minutes (over the relevant cortex area).
  Other Names: tDCS
  Arms: Crossover 1b: sham + anodal stimulation of M1
Device: Cathodal stimulation of M1 + sham — 8 active treatmments: 2mA cathodal stimulation of M1 for 20 minutes (over the relevant cortex area) , followed by 8 sham treatments.
  Other Names: tDCS
  Arms: Crossover 2a: cathodal stimulation of M1 + sham
Device: Sham + Cathodal stimulation of M1 — 8 sham treatments followed by 8 active treatmments: 2mA cathodal stimulation of M1 for 20 minutes (over the relevant cortex area).
  Other Names: tDCS
  Arms: Crossover 2b: sham + cathodal stimulation of M1

SUMMARY:
* Phantom limb pain (PLP) refers to pain in a limb that has been amputated or deafferented. Phantom limb pain might be related to brain cortical plastic changes.
* The purpose of this study is to determine the efficacy of a series of transcranial direct current stimulation (tDCS) sessions, a non-invasive and focal brain stimulation method, in producing long-term reduction of phantom limb pain among amputees who experience such pain.

This is a Crossover sham control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Limb amputation from at least 6 months before study enrollment
* Presence of PLP at least 2 times a week and present 4 weeks prior to onset of study
* Written informed consent

Exclusion Criteria:

* Coexistence of major neurological or psychiatric diseases
* Being actively enrolled in a separate study targeting pain relief
* Post traumatic stress disorder (PTSD) diagnosed patients
* Any contraindication to noninvasive brain stimulation such as past brain surgery, brain implants, cochlear implant, epilepsy or any past seizure
* Pregnant women
* Within the traumatic amputees group - subjects diagnosed with diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Reduced phantom limb pain | 5 months after last stimulation session
  Reduction of phantom limb pain compared to phantom limb pain before treatment, according to Visual Analog Scales (VAS) evaluation

SECONDARY OUTCOMES:
Adverse effects of treatment | Up to 5 weeks
  Severity of any adverse effects related to the transcranial direct current stimulation treatment will be checked after each stimulation session
Effects of treatment on the electrical activity of the brain | Up to 5 weeks
  Measurement of the electrical activity of the brain before, during and after each stimulation using an electroencephalography (EEG) device.

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Siev-Ner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Department of Orthopedic Rehabilitation, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Flor H. Phantom-limb pain: characteristics, causes, and treatment. Lancet Neurol. 2002 Jul;1(3):182-9. doi: 10.1016/s1474-4422(02)00074-1. PMID 12849487
- [Background] Cohen LG, Bandinelli S, Findley TW, Hallett M. Motor reorganization after upper limb amputation in man. A study with focal magnetic stimulation. Brain. 1991 Feb;114 ( Pt 1B):615-27. doi: 10.1093/brain/114.1.615. PMID 2004259
- [Background] Lotze M, Flor H, Grodd W, Larbig W, Birbaumer N. Phantom movements and pain. An fMRI study in upper limb amputees. Brain. 2001 Nov;124(Pt 11):2268-77. doi: 10.1093/brain/124.11.2268. PMID 11673327
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Nuti C, Peyron R, Garcia-Larrea L, Brunon J, Laurent B, Sindou M, Mertens P. Motor cortex stimulation for refractory neuropathic pain: four year outcome and predictors of efficacy. Pain. 2005 Nov;118(1-2):43-52. doi: 10.1016/j.pain.2005.07.020. Epub 2005 Oct 7. PMID 16214292
- [Background] Khedr EM, Ahmed MA, Fathy N, Rothwell JC. Therapeutic trial of repetitive transcranial magnetic stimulation after acute ischemic stroke. Neurology. 2005 Aug 9;65(3):466-8. doi: 10.1212/01.wnl.0000173067.84247.36. PMID 16087918
- [Background] Bolognini N, Olgiati E, Maravita A, Ferraro F, Fregni F. Motor and parietal cortex stimulation for phantom limb pain and sensations. Pain. 2013 Aug;154(8):1274-80. doi: 10.1016/j.pain.2013.03.040. Epub 2013 Apr 19. PMID 23707312
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] O'Connell NE, Cossar J, Marston L, Wand BM, Bunce D, Moseley GL, De Souza LH. Rethinking clinical trials of transcranial direct current stimulation: participant and assessor blinding is inadequate at intensities of 2mA. PLoS One. 2012;7(10):e47514. doi: 10.1371/journal.pone.0047514. Epub 2012 Oct 17. PMID 23082174
- [Background] Nitsche MA, Liebetanz D, Antal A, Lang N, Tergau F, Paulus W. Modulation of cortical excitability by weak direct current stimulation--technical, safety and functional aspects. Suppl Clin Neurophysiol. 2003;56:255-76. doi: 10.1016/s1567-424x(09)70230-2. No abstract available. PMID 14677403
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Kew JJ, Ridding MC, Rothwell JC, Passingham RE, Leigh PN, Sooriakumaran S, Frackowiak RS, Brooks DJ. Reorganization of cortical blood flow and transcranial magnetic stimulation maps in human subjects after upper limb amputation. J Neurophysiol. 1994 Nov;72(5):2517-24. doi: 10.1152/jn.1994.72.5.2517. PMID 7884476
- [Background] Chen R, Corwell B, Yaseen Z, Hallett M, Cohen LG. Mechanisms of cortical reorganization in lower-limb amputees. J Neurosci. 1998 May 1;18(9):3443-50. doi: 10.1523/JNEUROSCI.18-09-03443.1998. PMID 9547251
- [Background] Karl A, Birbaumer N, Lutzenberger W, Cohen LG, Flor H. Reorganization of motor and somatosensory cortex in upper extremity amputees with phantom limb pain. J Neurosci. 2001 May 15;21(10):3609-18. doi: 10.1523/JNEUROSCI.21-10-03609.2001. PMID 11331390
- [Background] Flor H, Elbert T, Knecht S, Wienbruch C, Pantev C, Birbaumer N, Larbig W, Taub E. Phantom-limb pain as a perceptual correlate of cortical reorganization following arm amputation. Nature. 1995 Jun 8;375(6531):482-4. doi: 10.1038/375482a0. PMID 7777055
- [Background] Roricht S, Meyer BU, Niehaus L, Brandt SA. Long-term reorganization of motor cortex outputs after arm amputation. Neurology. 1999 Jul 13;53(1):106-11. doi: 10.1212/wnl.53.1.106. PMID 10408544
- [Background] Yang TT, Gallen CC, Ramachandran VS, Cobb S, Schwartz BJ, Bloom FE. Noninvasive detection of cerebral plasticity in adult human somatosensory cortex. Neuroreport. 1994 Feb 24;5(6):701-4. doi: 10.1097/00001756-199402000-00010. PMID 8199341
- [Background] Hall EJ, Flament D, Fraser C, Lemon RN. Non-invasive brain stimulation reveals reorganized cortical outputs in amputees. Neurosci Lett. 1990 Aug 24;116(3):379-86. doi: 10.1016/0304-3940(90)90105-i. PMID 2243618
- [Background] Grusser SM, Winter C, Muhlnickel W, Denke C, Karl A, Villringer K, Flor H. The relationship of perceptual phenomena and cortical reorganization in upper extremity amputees. Neuroscience. 2001;102(2):263-72. doi: 10.1016/s0306-4522(00)00491-7. PMID 11166112
- [Background] Khedr EM, Kotb H, Kamel NF, Ahmed MA, Sadek R, Rothwell JC. Longlasting antalgic effects of daily sessions of repetitive transcranial magnetic stimulation in central and peripheral neuropathic pain. J Neurol Neurosurg Psychiatry. 2005 Jun;76(6):833-8. doi: 10.1136/jnnp.2004.055806. PMID 15897507
- [Background] Lefaucheur JP, Drouot X, Menard-Lefaucheur I, Zerah F, Bendib B, Cesaro P, Keravel Y, Nguyen JP. Neurogenic pain relief by repetitive transcranial magnetic cortical stimulation depends on the origin and the site of pain. J Neurol Neurosurg Psychiatry. 2004 Apr;75(4):612-6. doi: 10.1136/jnnp.2003.022236. PMID 15026508
- [Background] Brown JA, Barbaro NM. Motor cortex stimulation for central and neuropathic pain: current status. Pain. 2003 Aug;104(3):431-435. doi: 10.1016/S0304-3959(03)00209-4. No abstract available. PMID 12927615
- [Background] Fuhr P, Cohen LG, Dang N, Findley TW, Haghighi S, Oro J, Hallett M. Physiological analysis of motor reorganization following lower limb amputation. Electroencephalogr Clin Neurophysiol. 1992 Feb;85(1):53-60. doi: 10.1016/0168-5597(92)90102-h. PMID 1371745
- [Background] Elbert T, Sterr A, Flor H, Rockstroh B, Knecht S, Pantev C, Wienbruch C, Taub E. Input-increase and input-decrease types of cortical reorganization after upper extremity amputation in humans. Exp Brain Res. 1997 Oct;117(1):161-4. doi: 10.1007/s002210050210. PMID 9386015
- [Background] Birbaumer N, Lutzenberger W, Montoya P, Larbig W, Unertl K, Topfner S, Grodd W, Taub E, Flor H. Effects of regional anesthesia on phantom limb pain are mirrored in changes in cortical reorganization. J Neurosci. 1997 Jul 15;17(14):5503-8. doi: 10.1523/JNEUROSCI.17-14-05503.1997. PMID 9204932
- [Background] Tsubokawa T, Katayama Y, Yamamoto T, Hirayama T, Koyama S. Chronic motor cortex stimulation for the treatment of central pain. Acta Neurochir Suppl (Wien). 1991;52:137-9. doi: 10.1007/978-3-7091-9160-6_37. PMID 1792954
- [Background] Topper R, Foltys H, Meister IG, Sparing R, Boroojerdi B. Repetitive transcranial magnetic stimulation of the parietal cortex transiently ameliorates phantom limb pain-like syndrome. Clin Neurophysiol. 2003 Aug;114(8):1521-30. doi: 10.1016/s1388-2457(03)00117-2. PMID 12888036